CLINICAL TRIAL: NCT00852748
Title: Validation of Venogenic Hypothesis for Cough, Exertional and Sexual Headaches
Status: Completed | Type: Observational
Sponsor: French Society for the Study of Migraine Headache (Other)
Responsible Party: French Society for the Study of Migraine Headache, French Society for the Study of Migraine Headache
Other Study IDs: SFEMC 08.520
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2009-02

CONDITIONS: Headache
Keywords: headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical and neuroradiologic study concerning patients suffering of cough, exertional and sexual headaches disorders (pathophysiology) concerning a venous hypothesis implication, redescribe clinical headaches specifications, confirmed if cough headaches is a clinical entity and if it has neuroradiologic differences with effort or sexual activity headaches.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering of headache disorders

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering of cough, exertional and sexual headaches
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- assistance publique hopitaux de marseille CHU Timone, Marseille, France